CLINICAL TRIAL: NCT02156531
Title: An Efficacy-Effectiveness Trial of Cognitive Bias Modification for Youth Anxiety
Brief Title: Cognitive Bias Modification for Youth Anxiety
Acronym: TeenCBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01MH101118-01A1 (NIH); 1R01MH101118-01A1 (NIH)
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Anxiety
Keywords: Anxiety; Youth Anxiety; CBM; Cognitive Bias Modification; Adolescents
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Attention Control Condition (Placebo Comparator): 3.c.14.5. Arm 1: Attention Control Condition. The minimally effective attention-control group procedure is identical to the active CBM procedure except that during the presentation of the trials where a disgusted face is present, the probe will appear with equal frequency (50-50) in the position of disgusted or neutral face. Thus, the balanced (random) presentation of the probe in this condition is not designed to explicitly train attention away from threat and toward neutral stimuli, in contrast to the active versions of CBM in Arms 2 and 3.
  Interventions: Behavioral: Self-Administered, minimally effective attention-control version of the CBM program
- Arm 2: Self-administered CBM only (Experimental): 3.c.14.6. Arm 2: Self-Administered CBM Only. Youth assigned to this arm will receive the self-administered active CBM intervention. As described above in detail, in the 80% of CBM trials where a neutral and disgust face are both presented, the probe always replaces the neutral face. Thus, participants are trained to disengage their attention from threat. These youth do not receive Adherence Promotion telephone calls.
  Interventions: Behavioral: Self-Administered, Active Cognitive Bias Modification (CBM)
- Arm 3: Self-administered CBM + Adherence Promotion (Experimental): 3.c.14.7. Arm 3: Self-Administered CBM + Adherence Promotion. Youth assigned to this arm will receive both the self-administered active CBM intervention and the telephone coach calls to deliver the Adherence Promotion (AP) procedures. AP procedures are intended to compensate for the important nonspecific 'scaffolding' provided by research staff when CBM has been traditionally delivered in laboratories. This includes technical assistance with use of the program, support/encouragement, motivational enhancement, and brainstorming solutions to barriers to regular sessions. The addition of AP to the 3rd arm of this trial attempts to recreate much of this nonspecific, yet likely important, support of in-person interventions, which we hypothesize will lead to greater participant adherence to the program and therefore better clinical outcomes.
  Interventions: Behavioral: Self-Administered, Active Cognitive Bias Modification (CBM)

INTERVENTIONS:
Behavioral: Self-Administered, Active Cognitive Bias Modification (CBM) — Cognitive Bias Modification (CBM) is a novel treatment delivered via a downloadable computer program. CBM retrains individuals' attention away from negative/threatening stimuli and toward more balanced attention toward neutral stimuli.
  Arms: Arm 2: Self-administered CBM only; Arm 3: Self-administered CBM + Adherence Promotion
Behavioral: Self-Administered, minimally effective attention-control version of the CBM program — Identical to the active CBM program except that during the presentation of the trails where a disgusted face is present, the probe will appear with equal frequency (50-50) in the position of disgusted or neutral face. This, the balanced (random) presentation of the probe in this condition is not designed to explicitly train attention away from threat and toward neutral stimuli, in contrast to the active version of CBM.
  Arms: Attention Control Condition

SUMMARY:
Research in the last fifteen years suggests that anxious individuals selectively attend towards threatening information. Attention modification interventions for internalizing adults have been developed to target cognition at this basic level; these programs have demonstrated initial efficacy in attention bias and anxiety symptom reduction. To date, there have been minimal published studies of attention modification in youths with clinical levels of anxiety.

This study is a large randomized efficacy-effectiveness trial (N = 498) to test the benefit of this low-cost, computerized attention modification intervention (Cognitive Bias Modification (CBM) computer application) for anxiety disorders and symptomatology in youth ages 12 to 17. This trial conducted will compare three intervention arms, all of which include underlying treatment as usual (TAU). The investigators directly test the level of clinical support ("scaffolding") needed to adequately deliver self-administered CBM to anxious youth, a finding that will be key to preparing for future deployment-focused trials. The investigators will compare an attention control version of the CBM program (Arm 1) to two active versions of the CBM intervention that have varying levels of patient clinical support: a self-administered CBM program that participants download and install on their home computers (Self-Administered CBM-only; Arm 2), and the same CBM program paired with an adherence promotion (AP) component delivered via brief telephone calls from study "coaches," including as needed, brief motivational enhancement and/or technical assistance (Self-Administered CBM+AP; Arm 3).

The investigators expect that youth receiving CBM and CBM+AP will have improvement in anxiety symptoms and functioning. The investigators will also complete a cost-effectiveness analysis to examine potential costs offset by this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Youth age between 12.0 and 17.9 years old
* Youth, parent able to complete assessments in English
* Youth performing at 7th-12th grade achievement level
* Youth vision sufficient to read book of typical size print
* Youth access to home computer, Internet for 3 months
* Assessment of Childhood Disorders (ADIS)-confirmed diagnosis of generalized anxiety disorder (GAD) and/or social phobia (SOP) and/or separation anxiety disorder (SAD)

Exclusion Criteria:

* Youth diagnosis of learning or processing problem
* Youth diagnosis of attention deficit hyperactivity disorder (ADHD), except if symptoms are stable and controlled by medication for > 1 mo.
* Youth diagnosis of psychotic disorder
* Youth primary complaint of condition other than anxiety (as determined by the research interviewer during the baseline survey)
* psychotic features or delayed inform/visual processing

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2014-09; Primary Completion 2019-06 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness | 6 month follow up (post intervention)
  We hypothesize that CBM can be successfully delivered in this health-care setting, and that active CBM will demonstrate clinical effectiveness.
  Hypothesis 1a: The combined active CBM conditions will lead to greater rates of remission for anxiety diagnoses and to greater improvement on secondary indices of symptoms, diagnoses, and functioning, compared to the control condition (Arms 2 + 3 vs. Arm 1). Hypothesis 1b: CBM+AP will result in greater rates of remission for anxiety diagnoses (primary outcome) and greater improvement in secondary clinical indices, compared to CBM-only (Arm 3 vs. Arm 2).

SECONDARY OUTCOMES:
Cost Effectiveness | 12 months post intervention
  Overall, we expect that active CBM will be cost-effective from the healthcare organization perspective, including patient direct and indirect costs.
  Hypothesis 2a: Incremental cost-per-unit of anxiety-free-days (AFDs) and health-related quality of life (QALYS) will be lower for active CBM (Arm 2 + Arm 3), relative to the control condition (Arm 1) due to improvements in anxiety symptomology.
  Hypothesis 2b: Cost-per-unit of improved AFDs and QALYS will be lower in CBM-only (Arms 2) relative to CBM+AP (Arm 3). Although we expect both active CBM arms to improve anxiety, we expect that CBM+AP (Arm 3) will be considerably more costly due to increased labor costs of AP phone coaching, while producing only a moderate incremental clinical benefit beyond the effects of CBM only (Arm 2)

OTHER OUTCOMES:
Exploration of moderators associated with CBM effects | 12 months post intervention
  We will focus on moderators that may influence future dissemination, including whether CBM is robust to variation in youth clinical severity (e.g., baseline Clinical Global Impressions scale (CGI), severity of cognitive biases), comorbidity (e.g., depression), and demographics (e.g., gender, socioeconomic status, race/ethnicity). Our large sample allows for substantial variability on these characteristics.
Exploration of mediators associated with CBM effects | 12 months post intervention
  We will examine whether change in attentional bias mediates CBM effects and leads to improved anxiety, as posited by information-processing theories underlying the intervention.
Exploration of process variables associated with CBM effects | 12 months post intervention
  We will examine youth adherence to CBM, benchmarked against lab-based delivery of similar interventions (i.e., acceptable error rates) - this will include testing whether the CBM+AP condition results in higher participant engagement and compliance (e.g., high completion rates, low error rates) compared to conditions without AP (Arm 3 vs. Arms 1 + 2) and assessment of whether these process variables are associated with outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Clarke, PhD, Principal Investigator — Kaiser Permanente; Robin Weersing, PhD, Principal Investigator — San Diego State University; Nader Amir, PhD, Principal Investigator — San Diego State University
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Reetz S, Clarke G, Weersing R, Amir N, Dickerson J, Lynch FL, Leo MC, Rawlings AM, Lee MH, Gille S. The ReThink study: a 3-arm parallel randomized trial of cognitive bias modification, with and without adherence promotion, for adolescent anxiety disorder: trial design and protocol. BMC Psychiatry. 2019 Oct 22;19(1):306. doi: 10.1186/s12888-019-2296-z. PMID 31640613